CLINICAL TRIAL: NCT06273267
Title: Initial Pediatric Palliative Care Provision in Patients Under 25 Years of Age Classified in ACT Group 4 Within Ile de France (Metropolitan Area of Paris)
Brief Title: Initiating Pediatric Palliative Care in ACT Group 4
Acronym: StartSPP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231232
Record Dates: First submitted 2024-01-31; First posted 2024-02-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Encephalopathy; Cerebral Palsy; Cerebral Malformation; Traumatic Head Injury
Keywords: Serious incurable non-progressive neurological disease; Pediatric palliative care
MeSH Terms: conditions — Brain Diseases; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: AP-HP patients followed by the pediatric palliative care teams of Ile de France (metropolitan area of Paris) between January 2020 and December 2022 and suffering from a serious non-progressive neurological disease.
  Interventions: Other: Collection of data from the patient's medical file

INTERVENTIONS:
Other: Collection of data from the patient's medical file — Collection of data from the patient's medical file. The data collected concerns the first year of follow-up (from the initial PPC intervention to one year to date post-intervention).

SUMMARY:
Due to the wide range of diagnoses encountered in pediatric palliative care, the Association for Children's Palliative Care (ACT) and the Royal College of Paediatrics and Child Health (RCPCH) have developed a classification of life-limiting illnesses, based on support models.

This classification includes four groups. ACT 4 category is made up of children with a serious incurable non-progressive neurological disease (for example: anoxic ischemia, cerebral palsy, traumatic or infectious brain injuries).

Although data relating to specific ACT groups are scarce, experience from clinical practice suggests that the needs and use of Pediatric palliative care resources are different across the four categories.

The specific history of ACT-4 patients suggests that pediatric palliative care may be required early on in the history of the disease but effective intervention varies greatly from one patient to another. Tthis study aims to better understand the optimal timing for introducing a PPC team into the care pathway for these children. The study also aims to describe the care trajectory over the first year of PPC intervention.

DETAILED DESCRIPTION:
The ACT 4 group is made up of children with a serious incurable non-progressive neurological disease (for example: anoxic ischemia, cerebral palsy, traumatic or infectious brain injuries).

Although data relating to specific ACT groups are scarce, experience from clinical practice suggests that the needs and use of Pediatric palliative care resources are different across the four categories.

The question of when to initiate palliative care with curative pediatric care frequently arises for specialists in pediatrics and palliative medicine. In the ACT-4 group, where the pathologies are by definition non-progressive, the initial timing and mode of intervention of palliative care are less clear. The main reasons encountered in clinical practice are: symptomatic and therapeutic assessment, goals of care discussion, and implementing a care plan. Two main modes of intervention have been identified for hospital based teams (consultations and multidisciplinary meetings) and will be confirmed by extending the study to community care. The reasons and methods of intervention will be explored in our study.

The specific history of ACT-4 patients suggests that these patients may present pediatric palliative care needs early on, but effective intervention varies greatly from one patient to another. This study aims to better understand the optimal timing for introducing a PPC team into the care pathway for these children. The study also aims to describe the care trajectory over the first year of PPC intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 25
* Follow-ups at APHP
* Supported by a palliative care team from Ile de France (Robert-Debré hospital, Necker hospital or Paliped-Île-de-France Regional Pediatric Palliative Care Resource Team) between January 2020 and December 2022
* Suffering from a serious non-progressive neurological disease (ACT-4)
* Information and absence of opposition from the holders of parental authority of the minor patient and the guardian or curator of the adult patient if he is under guardianship/curatorship;

Exclusion Criteria:

* Other ACT category (1, 2, 3 or 5) of the classification of diseases by the Association for Children's Palliative Care (ACT) and the Royal College of Paediatrics and Child Health (RCPCH) during treatment
* Patients for whom there was no pediatric palliative care intervention
* Patients in palliative care without follow-up at the APHP

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: AP-HP (Assistance Publique - Hôpitaux de Paris) patients followed by the pediatric palliative care teams of the greater metropolitan area of Paris "Ile de France" (Robert-Debré hospital, Necker hospital or Paliped-Île-de-France Regional Pediatric Palliative Care Resource Team) between January 2020 and December 2022 and suffering from a serious non-progressive neurological disease.
  Robert Debré et Necker Hospitals are tertiary care hospitals. Paliped is a community based service for PPC.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Description of first pediatric palliative care intervention | 12 months
  The first pediatric palliative care team intervention will be listed for each patient (symptom management, multidisciplinary ethical meeting, care coordination, or team and family support). Collection of data from the patient's medical file. The data collected concerns the initial intervention.

SECONDARY OUTCOMES:
Description of the patient situation | 12 months
  Clinical description of the patient: ICD (international classification of diseases) diagnosis, acute symptoms, treatment, demographic characteristics and the place of care (hospital, hospice, palliative care unit, home).
  Collection of data from the patient's medical file. The data collected concerns the first year of follow-up, from the initial pediatric palliative care intervention to one year to date post-intervention.
Timing of pediatric palliative care intervention | 12 months
  Determine whether there is a significant difference in the reasons and modes of initiating pediatric palliative care depending on the precocity of the first intervention in relation to diagnosis and death if it has occurred. Analysis of time elapsed between diagnosis and palliative care intervention as well as time elapsed between palliative care and death if it has occured.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley RIDLEY, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris; Hélène GEFFROY, Resident, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Namisango E, Bristowe K, Allsop MJ, Murtagh FEM, Abas M, Higginson IJ, Downing J, Harding R. Symptoms and Concerns Among Children and Young People with Life-Limiting and Life-Threatening Conditions: A Systematic Review Highlighting Meaningful Health Outcomes. Patient. 2019 Feb;12(1):15-55. doi: 10.1007/s40271-018-0333-5. PMID 30361884
- [Background] Bender HU, Riester MB, Borasio GD, Fuhrer M. "Let's Bring Her Home First." Patient Characteristics and Place of Death in Specialized Pediatric Palliative Home Care. J Pain Symptom Manage. 2017 Aug;54(2):159-166. doi: 10.1016/j.jpainsymman.2017.04.006. Epub 2017 Jun 8. PMID 28602938
- [Background] DeCourcey DD, Silverman M, Oladunjoye A, Balkin EM, Wolfe J. Patterns of Care at the End of Life for Children and Young Adults with Life-Threatening Complex Chronic Conditions. J Pediatr. 2018 Feb;193:196-203.e2. doi: 10.1016/j.jpeds.2017.09.078. Epub 2017 Nov 22. PMID 29174080
- [Background] Good PD, Cavenagh J, Ravenscroft PJ. Survival after enrollment in an Australian palliative care program. J Pain Symptom Manage. 2004 Apr;27(4):310-5. doi: 10.1016/j.jpainsymman.2003.12.011. PMID 15050658
- [Background] Feudtner C, Kang TI, Hexem KR, Friedrichsdorf SJ, Osenga K, Siden H, Friebert SE, Hays RM, Dussel V, Wolfe J. Pediatric palliative care patients: a prospective multicenter cohort study. Pediatrics. 2011 Jun;127(6):1094-101. doi: 10.1542/peds.2010-3225. Epub 2011 May 9. PMID 21555495
- [Background] Siden H, Chavoshi N, Harvey B, Parker A, Miller T. Characteristics of a pediatric hospice palliative care program over 15 years. Pediatrics. 2014 Sep;134(3):e765-72. doi: 10.1542/peds.2014-0381. PMID 25157003
- [Background] Mack JW, Wolfe J. Early integration of pediatric palliative care: for some children, palliative care starts at diagnosis. Curr Opin Pediatr. 2006 Feb;18(1):10-4. doi: 10.1097/01.mop.0000193266.86129.47. PMID 16470155
- [Background] Himmelmann K, Sundh V. Survival with cerebral palsy over five decades in western Sweden. Dev Med Child Neurol. 2015 Aug;57(8):762-7. doi: 10.1111/dmcn.12718. Epub 2015 Feb 19. PMID 25694102